CLINICAL TRIAL: NCT05903157
Title: ME-WEL (MEnopause and WEight Loss): Protocol of a Randomised Controlled eHealth Intervention for Weight Management and Well-being in Post-Menopausal Women
Brief Title: ME-WEL: eHealth Behaviour Change Intervention for Weight Management in Post-menopausal Women
Acronym: ME-WEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SFRH/BD/144525/2019
Record Dates: First submitted 2023-05-25; First posted 2023-06-15 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Subjective Well-being; Weight Loss; Self Esteem; Physical Activity; Eating Behavior; Behavior and Behavior Mechanisms
MeSH Terms: conditions — Weight Loss; Motor Activity; Feeding Behavior; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Delivery of a health literacy flyer (Active Comparator): All Control Group participants received, through e-mail, a flyer about health literacy.
  Interventions: Behavioral: Control Group: Delivery of a health literacy flyer
- Weekly group sessions for weight management (Experimental): Participants in the Experimental Group were integrated into an eHealth 8-week group intervention, based on two theoretical models - the Health Action Process Approach (HAPA), and the Health Belief Model (HBM). Several Behaviour Change Techniques (BCT) were used, to promote the behaviour change.
  The experimental intervention consisted of: i) weekly group sessions (by Zoom platform), with a specific theme in each session, ii) weekly challenges, and iii) WhatsApp group interaction.
  Interventions: Behavioral: Experimental Group: Weekly group sessions for weight management

INTERVENTIONS:
Behavioral: Control Group: Delivery of a health literacy flyer — A health literacy flyer was delivered, by e-mail, in the first week of the intervention (the flyer contained its original source - the European Centre for Disease Prevention and Control). Beyond this, there was no further interaction with the group.
  All primary and secondary outcome measures were assessed at baseline, one month later (in the middle of the intervention), post-intervention, and follow-up moments (3 and 6 months after the intervention).
  Arms: Control Group: Delivery of a health literacy flyer
Behavioral: Experimental Group: Weekly group sessions for weight management — The eHealth intervention was designed based on: i) the Health Action Process Approach determinants, ii) the Health Belief Model constructs, and iii) behaviour change techniques (BCT, Taxonomy v1, by Michie et al., 2013) to implement healthy behaviours.
  The intervention consists of 8 sessions (90 minutes, once a week). All group intervention sessions, through the Zoom platform, are led by the psychologist responsible for the study. Whatsapp groups were created, to share experiences, knowledge, doubts, fears...
  All primary and secondary outcome measures were assessed at baseline, one month later (in the middle of the intervention), post-intervention, and in follow-up moments (3 and 6 months after the intervention).
  Arms: Weekly group sessions for weight management

SUMMARY:
In post-menopause, most women gain weight, and obesity rates are more prevalent in this particular group. In addition, there is an increased risk of cardiovascular disease, cancer, and diabetes. Given that this weight gain can be related to risk behaviours, healthy weight management (such as an increase in physical activity or healthy eating) is crucial to promote a healthy weight and well-being.

The ME-WEL (MEnopause and WEigth Loss) project (ref. SFRH/BD/144525/2019), entails an eHealth intervention for weight management and well-being in post-menopausal women with overweight or obesity, based on two theoretical models of behavioral change - the Health Action Process Approach (HAPA), and the Health Belief Model (HBM), and applying the Behaviour Change Techniques (BCT) Taxonomy and Oxford Food and Activity Behaviors (OxFAB) Taxonomy.

This group's eHealth intervention lasts 8 weeks. Each week there is a different theme to be addressed, taking into account the behavioral change models mechanisms, in articulation with different BCT´s and weight strategies.

Subjective well-being, self-esteem, weight loss, implementation of weight management strategies, and changes in eating behavior and physical activity/exercise were evaluated, through follow-ups at 3- and 6- post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age (45-65 years);
* Post-menopausal women (which starts after menopause/last period, confirmed by 12-month amenorrhea);
* Women with a Body Mass Index (BMI) of 25 kg/m2 or more (overweight) or women with a BMI of 30 kg/m2 or more (obesity);
* Nationality (Portuguese or dual nationality);

Exclusion Criteria:

* Specifical diseases and/or medical reasons to limit activity (stroke, cancer, diabetes, heart disease, epilepsy, musculoskeletal problems that severely compromise mobility; loss of functional ability);
* Diagnosis of mental health illness or recent hospitalization for mental health reasons;
* History of alcohol dependence;
* History of addiction to illicit substances;
* Suicidal ideation

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Positive and negative affect | Change from Baseline positive and negative affect one month after the intervention´s beginning, one week post-intervention, and at 3- and 6- months follow-ups
  Evaluated by "Short-Form of the Portuguese version of the positive and negative affect schedule - PANAS - Port - VRP" (Galinha et al., 2014)
Satisfaction with life scale | Change from Baseline satisfaction with life scale one month after the intervention´s beginning, one week post-intervention, and at 3- and 6- months follow-ups
  Evaluated by "Satisfaction with life scale" (Diener et al., 1985)
Weight management strategies | Change from Baseline weight management strategies one month after the intervention´s beginning, one week post-intervention, and at 3- and 6- months follow-ups
  Measured by the Oxford Food and Activity Behaviors Taxonomy (OxFAB-MAW; Leitão et al., 2023)

SECONDARY OUTCOMES:
Weight loss | Change from Baseline weight loss one month after the intervention´s beginning, one week post-intervention, and at 3- and 6- months follow-ups
  Assessed by Body Mass Index (BMI) - weight and height will be combined to report BMI in kg/m^2
Eating behaviour | Change from Baseline eating behaviour one month after the intervention´s beginning, one week post-intervention, and at 3- and 6- months follow-ups
  Measured by the Three Factor Eating Questionnaire (TFEQ-R21; Cappelleri et al., 2009)
Physical Activity | Change from Baseline physical activity one month after the intervention´s beginning, one week post-intervention, and at 3- and 6- months follow-ups
  Assessed by the International physical activity questionnaire (IPAQ; Craig et al., 2003)
Self-esteem | Change from Baseline self-esteem one month after the intervention´s beginning, one week post-intervention, and at 3- and 6- months follow-ups
  Assessed by the Rosenberg Self-Esteem Scale (RSS; Rosenberg, 1965)
Behaviour change (HAPA) | Change from Baseline behaviour change one month after the intervention´s beginning, one week post-intervention, and at 3- and 6- months follow-ups
  Assessed by HAPA Questionnaire (tailored to weight management), based on Godinho and collaborators' study (Godinho et al., 2014)
Behaviour change (HBM) | Change from Baseline behaviour change one month after the intervention´s beginning, one week post-intervention, and at 3- and 6- months follow-ups
  Evaluated by HBM questionnaire (tailored to weight management), based on Saghafi-Asl and collaborators' study (2020).

CONTACTS AND LOCATIONS:
Overall Officials: Filipa Pimenta, Ph.D., Study Chair — WJCR, Ispa - Instituto Universitário
Locations (1):
- Ispa - Instituto Universitário, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Background] Leitao M, Hartmann-Boyce J, Perez-Lopez FR, Maroco J, Pimenta F. Weight management strategies in Middle-Aged Women (MAW): Development and validation of a questionnaire based on the Oxford Food and Activity Behaviors Taxonomy (OxFAB-MAW) in a Portuguese sample. Front Psychol. 2023 Jan 4;13:1069775. doi: 10.3389/fpsyg.2022.1069775. eCollection 2022. PMID 36687937
- [Background] Godinho CA, Alvarez MJ, Lima ML, Schwarzer R. Will is not enough: coping planning and action control as mediators in the prediction of fruit and vegetable intake. Br J Health Psychol. 2014 Nov;19(4):856-70. doi: 10.1111/bjhp.12084. Epub 2013 Dec 6. PMID 24308823
- [Background] Saghafi-Asl M, Aliasgharzadeh S, Asghari-Jafarabadi M. Correction: Factors influencing weight management behavior among college students: An application of the Health Belief Model. PLoS One. 2021 May 20;16(5):e0252258. doi: 10.1371/journal.pone.0252258. eCollection 2021. PMID 34015038